CLINICAL TRIAL: NCT02941380
Title: Cerebral Oxidative and Inflammatory Stress and Cerebral Hemodynamics During and After Coronary Artery Bypass Grafting With Use of Cardiopulmonary Bypass
Brief Title: Exploration of Cerebral Pathophysiology During and After CABG Using CPB
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Claus Behrend Christiansen, M.D., Rigshospitalet, Denmark
Other Study IDs: H-4-2011-037
Record Dates: First submitted 2016-04-29; First posted 2016-10-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Ischemic Heart Disease
Keywords: coronary artery bypass grafting; cardiopulmonary bypass; Cerebral oxidative stress; Cerebral inflammatory stress; Cerebral hemodynamics; Postoperative cognitive dysfunction
MeSH Terms: conditions — Myocardial Ischemia; Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ischemic heart disease: Patients admitted for coronary artery bypass grafting with the use of cardiopulmonary bypass

SUMMARY:
Purpose:

The purpose of this study is to examine cerebral oxidative and inflammatory stress and cerebral hemodynamics during and after coronary artery bypass grafting and correlate with postoperative cognitive function.

DETAILED DESCRIPTION:
Postoperative cognitive decline is a well-known and well-described complication following coronary artery bypass grafting. Severity ranges from postoperative delirium to stroke, but the majority of patients with postoperative cognitive decline following coronary artery bypass grafting have decline in recent and remote memory in particular.

The reason for the cognitive decline is still not fully understood though many reasons have been proposed.

Inflammation and oxidative stress may contribute to the postoperative cognitive dysfunction which may also be in combination with a reduced cerebral autoregulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic heart disease admitted for coronary artery bypass grafting with the use of cardiopulmonary bypass

Exclusion Criteria:

* Cerebrovascular disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic heart disease admitted for coronary artery bypass grafting with the use of cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Cerebral autoregulation | 6 hours post operation
  Flow measurement of middle cerebral artery and measurement of middel arterial pressure

SECONDARY OUTCOMES:
Postoperative cognitive function | One day prior to operation and three days after operation

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Møller, MD PhD DMSc, Study Director — Rigshospitalet, Denmark

IPD SHARING:
Plan to Share IPD: No